CLINICAL TRIAL: NCT07126418
Title: Sex-Based Differences in Cervical Joint Position Sense and Disability in Patients With Chronic Mechanical Neck Pain: A Cross-Sectional Study
Brief Title: Sex-Based Differences in Cervical Joint Position Sense in Patients With Chronic Mechanical Neck Pain
Status: Completed | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Hoda Ibrahim Abbas Mousa, Principal Investigator, Cairo University
Other Study IDs: P.T.REC/012/003940; P.T.REC/012/006048 (Other: Faculty of physical therapy research ethical committee)
Record Dates: First submitted 2025-08-10; First posted 2025-08-17 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Chronic Mechanical Neck Pain
MeSH Terms: interventions — Observation

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- group A:30 males' patients with a primary complaint of chronic neck pain more than 3 months
  Interventions: Other: observation (cervical proprioception, neck pain and neck disability)
- Group B: 30 females' patients with a primary complaint of chronic neck pain more than 3 months
  Interventions: Other: observation (cervical proprioception, neck pain and neck disability)

INTERVENTIONS:
Other: observation (cervical proprioception, neck pain and neck disability) — 1) Assessment of cervical proprioception using CROM device: Head reposition accuracy tests: neutral head position (NHP) and target head position (THP) tests are common tests used to assess cervical proprioception. Repositioning to the NHP and repositioning into THP. The test procedures were the same as those described by Lee et al., 2006. The NHP test measures the subject's ability to actively reposition their head to their self-selected neutral position. The THP test measures the individual's ability to actively reposition the head to a previously demonstrated target position. A) Neutral head position: After explaining the testing procedure, the CROM device will securely fixed on the head of the subject. The participants will instructed to sit upright with their feet flat on the floor, their back against the chair backrest and facing straight ahead, this position will established as their self-selected "NHP".
  The magnetic part of the unit was then placed so that it was put

SUMMARY:
This is across sectional observational study aims to investigate whether there are sex-based differences in cervical proprioception, pain intensity, and neck disability in patients with chronic mechanical neck pain. The findings may contribute to better individualized care plans and inform future clinical guidelines.

DETAILED DESCRIPTION:
Neck pain is a common condition and one of the leading causes of disability worldwide, with mean estimates of 7.6% point prevalence (range, 5.9-38.7%), 37% annual prevalence (range, 16.7-75%), and 48.5% lifetime prevalence(range, 14.2-71%).

Although neck pain can be attributed to traumatic (such as whiplash associated) disorders, metabolic, neoplastic, inflammatory, or infectious diseases, most neck pain has no discernable cause and is considered to be idiopathic.

Chronic mechanical neck pain (CMNP) is a prevalent musculoskeletal condition, particularly among working-age adults, with a higher prevalence observed in females compared to males. The condition is commonly associated with impairments in cervical proprioception, pain, and functional disability. Cervical joint position sense (JPS) is a crucial component of sensorimotor control and has been found to be impaired in individuals with chronic neck pain.

The clinical practice guidelines for chronic idiopathic neck pain do not support percutaneous or open surgical treatment and recommend conservative treatment. However, as conservative treatment usually fails to maintain long-term efficacy, clinical studies begin to pay attention to the evaluation and management of proprioceptive dysfunction in patients with idiopathic neck pain.

Sex differences in pain perception and musculoskeletal disorders have been well-documented in the literature. A previous study revealed that the repositioning accuracy of the knee joint was significantly lower in female participants than in males and Sex-based difference in the accuracy of knee joint proprioception may imply that knee proprioceptive sensitivity might potentially contribute to the high incidence of knee injury in females compared with males. Another study showed that shoulder position sense, as part of the neuromuscular control system, differs between men and women. the findings showed a significant difference in constant position sense error between men and women and a significantly higher variability in the performance of men compared to women.

However, limited studies have directly compared cervical proprioception between males and females in the context of chronic mechanical neck pain. Understanding these differences is essential for optimizing rehabilitation strategies and personalizing interventions.

This study aims to investigate whether there are sex-based differences in cervical proprioception, pain intensity, and neck disability in patients with chronic mechanical neck pain. The findings may contribute to better individualized care plans and inform future clinical guidelines.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a primary complaint of chronic neck pain (assessed by VAS )for more than 3 months .
* patients with age range from 18 to 45 years old.
* patients with body mass index less than 30 kg/m2

Exclusion Criteria:

* previous spine surgery
* pregnancy.
* Diabetic patients
* Hypertensive patients
* Patients were excluded if neck pain was associated with cervical radiculopathy, whiplash injuries or severe headaches -cervical spine fracture - vertebrobasilar insufficiency.
* red flags suggesting of cancer, infection, vascular insufficiency
* Rheumatologic condition as mild systemic lupus erythematosus, poly-articular osteoarthritis, rheumatoid arthritis and advanced cervical spine degenerative diseases.
* patients received any form of cervical treatments within past 6 months

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: * Sixty patients 30 males and 30 females (diagnosed and referred from orthopedist ) with a primary complaint of chronic neck more than 3 months, will be selected .
  * All subjects will participate in the study after signing institutionally approved consent form prior to data collection.
Sampling Method: Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2025-09-10 (Actual); Primary Completion 2026-02-01 (Actual); Study Completion 2026-02-01 (Actual)

PRIMARY OUTCOMES:
cervical joint position Error (JPE) measured with CROM device at baseline | at baseline

SECONDARY OUTCOMES:
pain intensity: Visual Analog Scale (VAS) will be used to assess pain intensity at baseline | at baseline
  . Scores are based on self-reported measures of symptoms that are recorded with a single handwritten mark placed at one point along the length of a 10-cm line that represents a continuum between the two ends of the scale- "no pain" on the left end (0 cm) of the scale and the "worst pain" on the right end of the scale (10 cm)
Dysfunction of neck area: The neck disability index (NDI) will used to assess the level of cervical dysfunction | at baseline
  It is a patient-completed, condition-specific functional status questionnaire with 10 items.The NDI can be scored as a raw score or doubled and expressed as a percent. Each section is scored on a 0 to 5 rating scale, in which zero means 'No pain' and 5 means 'Worst imaginable pain'. Al the points can be summed to a total score. The test can be interpreted as a raw score, with a maximum score of 50, or as a percentage. 0 points or 0% means: no activity limitations, 50 points or 100% means complete activity limitation. A higher score indicates more patient-rated disability

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo University- Faculty of physical therapy, Cairo, Egypt